CLINICAL TRIAL: NCT00051428
Title: The Efficacy of Reiki in the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001075-01 (NIH)
Record Dates: First submitted 2003-01-09; First posted 2003-01-15 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia, Reiki, Energy Medicine
MeSH Terms: conditions — Fibromyalgia | interventions — Therapeutic Touch

INTERVENTIONS:
Procedure: Reiki (distant and direct-contact)

SUMMARY:
The purpose of this study is to investigate the effectiveness of Reiki in the treatment of fibromyalgia (FM), a condition characterized by widespread muscle pain and stiffness, often accompanied by sleep disturbance, headaches, irritable bowel syndrome, and psychological distress. Reiki is a form of energy medicine in which practitioners reportedly access universal life energy to heal patients, either by direct contact at specific hand positions or from a distance.

DETAILED DESCRIPTION:
Fibromyalgia is one of the most common rheumatologic diagnoses. Treatment is generally unsatisfactory and most randomized, controlled treatment trials have been unable to demonstrate a sustained effective intervention. A vast body of anecdotal literature as well as two randomized controlled trials suggest that Reiki may be an effective treatment for FM, appearing to relieve pain and improve psychological well being. Reiki appears to have no adverse effects and can eventually be self-administered, making it a low-risk, low-cost, potentially patient-empowering intervention. This study will investigate the efficacy of Reiki in the treatment of FM.

One hundred Reiki-naive FM patients will be recruited from a chronic fatigue referral clinic and will participate in an 8-week trial. Patients will be randomized into one of two Reiki groups (direct-contact and distant Reiki) or one of two control groups (sham and placebo). Patients will receive either Reiki or placebo 16 times during the course of the study. Patients will be assessed at study entry, at Weeks 4 and 8, and 12 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria

* Fibromyalgia without concurrent medical conditions associated with chronic pain, such as diabetic neuropathy, systemic lupus erythematosus, or severe degenerative joint disease
* Willing to undergo randomization and attend treatments regularly
* Willing to stay on a stable medical regimen during the entire 8-week trial and use only acetaminophen for breakthrough pain
* Live within a one-hour drive of the study site

Exclusion Criteria

* Received Reiki or any other energy medicine (Therapeutic Touch, Qi Gong, SHEN Therapy, etc.)
* Pregnant
* Pending litigation or disability claim related to FM

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-01; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Dedra S. Buchwald, Principal Investigator — University of Washington
Locations (1):
- Univ of WA - CFS/FM Research Center, Seattle, Washington, United States